CLINICAL TRIAL: NCT03984292
Title: Development of Laparoscopic Skills in Medical Students - What Makes the Difference?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Rizwan Khan, Associate Professor of Surgery, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 172008SUR
Record Dates: First submitted 2019-05-26; First posted 2019-06-12 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Clinical Skills

STUDY DESIGN:
Intervention Model Description: The students will be randomly distributed into two groups by using pre-designed envelopes:
  Group I: Single teaching session of 3 hours at single encounter Group II: 3 teaching sessions of 1 hour each over a period of 3 weeks The study will be open to all the year 2, 3 and 4 medical students of Aga Khan University Medical College and recruitment shall be done on first come-first serve basis.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor shall not be aware of the type of training which has been given to the students.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mass Learning (Experimental): Single teaching session of 3 hours shall be provided
  Interventions: Procedure: Teaching of laparoscopic skills on a box simulator
- Distributed Learning (Experimental): Three teaching sessions of 1 hour each shall be provided.
  Interventions: Procedure: Teaching of laparoscopic skills on a box simulator

INTERVENTIONS:
Procedure: Teaching of laparoscopic skills on a box simulator — The students shall be trained a laparoscopic simulator for a variable duration and the outcome shall be compared.

SUMMARY:
Learning is a complex process and influenced by a number of factors including the innate ability of the trainee, previous experiences (e.g. video game skills, music instrument skills), learning style and the overall learning environment. Understanding of the learning process and factors influencing the learning shall help develop and plan an effective curriculum for the trainees.

The investigators plan to use medical students as a part of the study since they have little or no prior knowledge or experience of laparoscopic skills. If any factors are identified, the investigators can help guide the participants for future training as well as develop a comprehensive curriculum for the current surgical trainees.

The primary objective of the study is to determine if acquisition and retention of laparoscopic skills in medical students is superior with multiple training sessions as compared to a single training session of the similar duration.

DETAILED DESCRIPTION:
Study Design:

This will be a parallel randomised controlled study design with a 1:1 ratio in each arm studying the influence of duration and number of training encounters on the acquisition of laparoscopic surgery skills.

Setting: The training shall be conducted at the Centre for Innovation in Medical Education (CIME) of the Aga Khan University, Karachi, Pakistan. The data shall be collected and analysed at the department of surgery of Aga Khan University, Karachi, Pakistan.

Study Participants: Year 2, 3 and 4 medical students of Aga Khan University Medical College, Karachi, will be invited to voluntarily participate in the study.

Sample Size & Groups: A non-probability, all-inclusive sampling technique will be used. A voluntary participation will be required and the expected number of participants has been estimated to be 50 in each group. The students will be randomly distributed into two groups by using pre-designed envelopes:

Group I: Single teaching session of 3 hours at single encounter Group II: 3 teaching sessions of 1 hour each over a period of 3 weeks The study will be open to all the year 2, 3 and 4 medical students of Aga Khan University Medical College and recruitment shall be done on first come-first serve basis. The sample size of 50 has been calculated based on the convenience using the data from previous studies. The usual class at AKU consists of 100 students and it is expected that at least 33% would consent to participate in the study. There are no specific exclusion criteria for this group of medical students.

Intervention: The intervention will be based on training sessions of 15-minute tutorial on basic principles of instrument handling, depth perception and hand eye coordination followed by live demonstration of specific tasks. This will be followed by hands-on practice by the participants of the following tasks:

1. Transfer of pegs / bean balls across dishes by non-dominant hand
2. Passing thread through hooks using dominant hand
3. Precision cutting - cutting a circle on gauze / paper with endo-scissors The participants in each arm will be further sub-divided in a group of 10 and each sub-group will be facilitated by a designated general surgeon who is expert in laparoscopic skills.

For group I, there will be 'one' training session lasting for 3 hours. For group II, the training shall consist of 'three' sessions of one hour each distributed over a period of 3 weeks. Hence the total duration of training will be the same in both groups, but the period of learning shall be different.

Outcome Assessment:

1. Baseline Assessment: At the initial encounter, an informed consent shall be taken from the medical students and they will be asked to complete a questionnaire describing their demographics, dominant hand, interest in future specialty and hobbies including playing video games and musical instruments. This will be followed by assessment of baseline psychomotor skills of the participants on laboratory-based models (described below). The skills assessed will focus on use of dominant hand, depth perception, and hand-eye coordination.
2. Pre- and Post-intervention Assessment: The participants shall be asked to complete the specific tasks described above before and after the intervention. The performance shall be monitored by the designated supervising faculty with expertise in laparoscopic skills and graded in terms of efficiency and quality of performance. The scale used to grade the students' skills will be the previously validated scale for assessment of laparoscopic skills known as GOALS (Global assessment of laparoscopic skills)21. Each participant shall be given 300 seconds to complete each task with negative marking for any deviation. Pre-intervention assessment shall be performed immediately before the training for both the groups while post-intervention assessment shall be performed at the completion of total duration of training for each group i.e. immediate for group I and at 3 weeks for group II.
3. Interval Assessment: All the participants will be scheduled for interval assessment of their skills at 3 months, 6 months and 1-year after the intervention. It is expected that the students shall not undergo any formal training in laparoscopic skills since this is not a part of their curriculum, but they can continue with their hobbies. The rationale behind this on-going assessment is to monitor longitudinal retention of knowledge after short learning encounters.

Assessment of Performance: Actual content and duration of training of the two groups shall be similar except that one group shall have a single session of mass training while the second group shall have 3 sessions of distributed practice. The technical skills of the students shall be assessed by the surgeons experienced in laparoscopic surgery as well as assessment of performance of medical students. The surgeon performing the assessment before and after the intervention shall be blinded to the type of training offered to the students. The assessment will be objective in terms of time duration taken to complete the task with negative marking for any deviation. If student is unable to complete the task during the given time frame, additional time required to complete the task shall be calculated based on the actual part of the task completed.

Randomization: The students in each arm will be randomized by using the pre-designed envelopes. The selection of students, development of blinded envelopes and randomization will be done by the primary investigator. The facilitating faculty shall be aware of the randomization for each group, but the assessing faculty shall be kept blinded to this randomization.

Statistical Analysis: Demographic data and distribution of hobbies will be described in frequencies and percentage. The scores at various readings will be described as mean, median, minimum and maximum values with standard deviations. The pre-intervention, post-intervention and interval assessment mean scores will be compared by using repeat measures of ANOVA. The effect of gender and hobbies on the scores will be analyzed by using one way ANOVA. The level of significance will at 0.05.

Ethical Clearance: An ethical approval for the conduct of the study will be obtained from the institutional ethics committee. An informed consent will be obtained from the participants for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical students of years 2, 3 and 4 with interest in laparoscopic surgery skills who volunteer to participate in the study

Exclusion Criteria:

* The students who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical Skills | 1 year
  Clinical skills of students shall be assessed by using the GOALS (global operative assessment of laparoscopic skills) scale for assessment of clinical skills in laparoscopy. This is a validated tool and has 5 parameters assessed on a Likert scale of 1 to 5. Higher the score, better the value.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Rizwan Khan, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual data not to be shared